CLINICAL TRIAL: NCT07086690
Title: Comparative Evaluation of Nebulized Ketamine, Nebulized Combination of Ketamine and Dexmedetomidine and Intramuscular Ketamine for Procedural Sedation and Analgesia in Pediatric Burn Injuries
Brief Title: Comparing Nebulized Ketamine,Nebulized Ketamine and Precedex and IM Ketamine for Analgesia in Pediatric Burn
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MD89/2025
Record Dates: First submitted 2025-05-21; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-04

CONDITIONS: Inhalation Anesthesia
MeSH Terms: interventions — Population Groups; Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients will receive nebulized ketamine (Active Comparator): Group (1): Patients will receive nebulized ketamine (2 mg/kg) Drugs will be prepared in 3 mL of saline 0.9% before administration by a standard hospital jet nebulizer via a mouthpiece, with a continuous flow of oxygen at 6 L/min for 10 to 15 minutes. Treatment will be stopped when the nebulizer begin to sputter. All solutions will be prepared in identical syringes with matching random codes by an independent investigator not involved in the observation or the administration of the anesthesia.
  Interventions: Drug: Group (1): Patients will receive nebulized ketamine (2 mg/kg)
- Group (2): Patients will receive nebulized combination of dexmedetomidine and ketamine (1 μg/kg + 1 (Active Comparator): Group (2): Patients will receive nebulized combination of dexmedetomidine and ketamine (1 μg/kg + 1 mg/kg) Drugs will be prepared in 3 mL of saline 0.9% before administration by a standard hospital jet nebulizer via a mouthpiece, with a continuous flow of oxygen at 6 L/min for 10 to 15 minutes. Treatment will be stopped when the nebulizer begin to sputter. All solutions will be prepared in identical syringes with matching random codes by an independent investigator not involved in the observation or the administration of the anesthesia.
  Interventions: Drug: Group (2): Patients will receive nebulized combination of dexmedetomidine and ketamine (1 μg/kg + 1 mg/kg)
- - Group (3): Patients will receive intramuscular ketamine (4 mg/kg, intramuscularly) 15 mins before (Active Comparator): - Group (3): Patients will receive intramuscular ketamine (4 mg/kg, intramuscularly) 15 mins before starting the procedure.
  Drugs will be prepared in 3 mL of saline 0.9% before administration by a standard hospital jet nebulizer via a mouthpiece, with a continuous flow of oxygen at 6 L/min for 10 to 15 minutes. Treatment will be stopped when the nebulizer begin to sputter. All solutions will be prepared in identical syringes with matching random codes by an independent investigator not involved in the observation or the administration of the anesthesia.
  Interventions: Drug: Patients will receive intramuscular ketamine (4 mg/kg, intramuscularly) 15 mins before starting the procedure.

INTERVENTIONS:
Drug: Group (1): Patients will receive nebulized ketamine (2 mg/kg) — Drugs will be prepared in 3 mL of saline 0.9% before administration by a standard hospital jet nebulizer via a mouthpiece, with a continuous flow of oxygen at 6 L/min for 10 to 15 minutes. Treatment will be stopped when the nebulizer begin to sputter. All solutions will be prepared in identical syringes with matching random codes by an independent investigator not involved in the observation or the administration of the anesthesia.
  - All patients will be admitted on the day of the surgery and will be instructed to fast 6 hours before surgery for older patients, as for breast fed patients, they will be instructed for 4 hours for breast feeding and for formula fed patients they will be instructed to fast for 6 hours as recommended by the American society of anesthesiologists. Preoperative assessment will be done before surgery by one of the members of the team who will make sure that the inclusion and exclusion criteria of the patients are considered, and baseline vital signs willbe rec
  Other Names: Not present
  Arms: Patients will receive nebulized ketamine
Drug: Group (2): Patients will receive nebulized combination of dexmedetomidine and ketamine (1 μg/kg + 1 mg/kg) — Drugs will be prepared in 3 mL of saline 0.9% before administration by a standard hospital jet nebulizer via a mouthpiece, with a continuous flow of oxygen at 6 L/min for 10 to 15 minutes. Treatment will be stopped when the nebulizer begin to sputter. All solutions will be prepared in identical syringes with matching random codes by an independent investigator not involved in the observation or the administration of the anesthesia.
  - All patients will be admitted on the day of the surgery and will be instructed to fast 6 hours before surgery for older patients, as for breast fed patients, they will be instructed for 4 hours for breast feeding and for formula fed patients they will be instructed to fast for 6 hours as recommended by the American society of anesthesiologists. Preoperative assessment will be done before surgery by one of the members of the team who will make sure that the inclusion and exclusion criteria of the patients are considered, and baseline vital signs will be re
  Other Names: Nebulized ketamine and precedex
  Arms: Group (2): Patients will receive nebulized combination of dexmedetomidine and ketamine (1 μg/kg + 1
Drug: Patients will receive intramuscular ketamine (4 mg/kg, intramuscularly) 15 mins before starting the procedure. — Drugs will be prepared in 3 mL of saline 0.9% before administration by a standard hospital jet nebulizer via a mouthpiece, with a continuous flow of oxygen at 6 L/min for 10 to 15 minutes. Treatment will be stopped when the nebulizer begin to sputter. All solutions will be prepared in identical syringes with matching random codes by an independent investigator not involved in the observation or the administration of the anesthesia.
  - All patients will be admitted on the day of the surgery and will be instructed to fast 6 hours before surgery for older patients, as for breast fed patients, they will be instructed for 4 hours for breast feeding and for formula fed patients they will be instructed to fast for 6 hours as recommended by the American society of anesthesiologists. Preoperative assessment will be done before surgery by one of the members of the team who will make sure that the inclusion and exclusion criteria of the patients are considered, and baseline vital signs will be re
  Other Names: Not present
  Arms: - Group (3): Patients will receive intramuscular ketamine (4 mg/kg, intramuscularly) 15 mins before

SUMMARY:
The present study compares efficacy of nebulised ketamine and combination of nebulised dexmedetomidine and ketamine and intramuscular ketamine for procedural sedation and analgesia in pediatric burn injuries

DETAILED DESCRIPTION:
Written informed consent will be obtained from parents of all participants prior to the study.

* Demographic information (age, sex, ethnicity).
* Clinical history and physical examination (Heart rate, Hypertension, Respiratory rate, burn percentage …. etc).
* Intervention:

  * Group (1): Patients will receive nebulized ketamine (2 mg/kg)
  * Group (2): Patients will receive nebulized combination of dexmedetomidine and ketamine (1 μg/kg + 1 mg/kg) Drugs will be prepared in 3 mL of saline 0.9% before administration by a standard hospital jet nebulizer via a mouthpiece, with a continuous flow of oxygen at 6 L/min for 10 to 15 minutes. Treatment will be stopped when the nebulizer begin to sputter. All solutions will be prepared in identical syringes with matching random codes by an independent investigator not involved in the observation or the administration of the anesthesia.
* Group (3): Patients will receive intramuscular ketamine (4 mg/kg, intramuscularly) 15 mins before starting the procedure. (Green et al., 1998).
* All patients will be admitted on the day of the surgery and will be instructed to fast 6 hours before surgery for older patients, as for breast fed patients, they will be instructed for 4 hours for breast feeding and for formula fed patients they will be instructed to fast for 6 hours as recommended by the American society of anesthesiologists. Preoperative assessment will be done before surgery by one of the members of the team who will make sure that the inclusion and exclusion criteria of the patients are considered, and baseline vital signs will be recorded. According to randomization that will be done by a computerized program, the drug will be administered to the patients in the preparation room by a researcher who will not participate in the evaluation of the patients before transfer to the operation room (OR).
* Parents are not allowed to accompany their children to the OR according to the hospital policy.
* Upon arrival to the OR department the Parental separation anxiety scale (PSAS) will be calculated.

Upon entering the operation room, standard monitoring will be commenced including ECG, non-invasive blood pressure and pulse oximetry and baseline measurement will be recorded. An attempt of cannulation will be done by an expert.

* During the length of the operation vital data will be recorded at 5 minutes interval. all patients will receive IV paracetamol 15mg/kg and patient would receive 3 mg/kg propofol as a rescue dose if vital data increased by >20% of the baseline. Sedation will be assessed by University of Michigan Sedation Scale (UMSS) After the completion of procedure, patient will be discharged to post-anesthesia care unit (PACU) in for the first 15 min. During the stay in PACU pain will also be assessed by using FLACC score.
* Discharge from PACU will be done after meeting discharge criteria and the time of discharge will be documented. After discharge pain score will be measured using FLACC score at 15, 30, 60 minutes interval postoperative and the total combustion of postoperative analgesics will be calculated as well as the time of discharge from the hospital

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologists (ASA) physical status I & II
* Pediatrics aged from 3 to 10 years.
* Both genders
* Pediatrics that has burn injuries and need sedation for cannulation and dressing.
* Burn >5% body surface area and <20% of surface area

Exclusion Criteria:

* ASA III and V patients with history of chronic illness
* Patients with known allergy/hypersensitivity to the study drug
* Congenital diseases or developmental delay or with neurological disease,
* known case of bronchial asthma or difficult airway were excluded from the study
* parents' refusal for participation in the study
* Emergency surgeries with hemodynamic instability
* mental retardation,
* neurological or psychiatric illness that may be associated with anxiety and agitation (cerebral palsy, seizure, separation anxiety disorder, ADHD etc.).
* treatment with anticonvulsants and sedatives
* Major sepsis or extensive infection

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2027-04-16 (Estimated); Study Completion 2027-04-16 (Estimated)

PRIMARY OUTCOMES:
Comparative evaluation of nebulized ketamine, nebulized combination of ketamine and dexmedetomidine and intramuscular ketamine for procedural sedation and analgesia in pediatric burn injuries | 5 minutes
  * The primary outcome will be depth of sedation evaluated by (UMSS) upon transfer to OR (after patient separation)
  * During the length of the operation vital data will be recorded at 5 minutes interval. all patients will receive IV paracetamol 15mg/kg and patient would receive 3 mg/kg propofol as a rescue dose if vital data increased by >20% of the baseline. Sedation will be assessed by University of Michigan Sedation Scale (UMSS) Value Patient state 0 Awake and alert
  Minimally sedated: tired/sleepy, appropriate response to verbal conversation, and/or sound 2 Moderately sedated: somnolent/sleeping, easily aroused with light tactile stimulation or a simple verbal command 3 Deeply sedated: deep sleep, aroused only with significant physical stimulation 4 Unarousable

SECONDARY OUTCOMES:
Comparative evaluation of nebulized ketamine, nebulized combination of ketamine and dexmedetomidine and intramuscular ketamine for procedural sedation and analgesia in pediatric burn injuries | 1 hour
  * analgesic effect using FLACC
  * After the completion of procedure, patient will be discharged to post-anesthesia care unit (PACU) in for the first 15 min. During the stay in PACU pain will also be assessed by using FLACC score:
  Behavior 0
  1 Face No particular expression or smile Occasional grimace or frown, withdrawn, disinterested Legs Normal position or relaxed Uneasy, restless, tense Activity Lying quietly, normal position, moves easily Squirming, shifting, back and forth, tense Cry No cry (awake or asleep) Moans or whimpers; occasional complaint Consolability Content, relaxed Reassured by touching, hugging, or being talked to, distractible

OTHER OUTCOMES:
Parental seperation anxiety scale | 10 minutes
  - Upon arrival to the OR department the Parental separation anxiety scale (PSAS) will be calculated according to the following: Behavior of the child during separation from parents Criteria score Excellent Patient unafraid, cooperative, or asleep
  1 Good Slightly afraid/crying, quiet with reassurance 2 Fair Moderately afraid and crying not quit with reassurance 3 Poor Crying, need for restraint 4
Recovery time | 1 hour
  How long will the patient need to be fully conscious

CONTACTS AND LOCATIONS:
Overall Officials: Marihan A Lwiz, MBBCH,M.Sc., Principal Investigator — Teaching assistant Ain Shams university
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1/2028
Access Criteria: Free